## Statistical Analysis Plan Final Analysis

A DOUBLE-BLIND PLACEBO CONTROLLED RANDOMIZED PHASE III TRIAL OF FULVESTRANT AND IPATASERTIB AS TREATMENT FOR ADVANCED HER-2 NEGATIVE AND ESTROGEN RECEPTOR POSITIVE (ER+) BREAST CANCER FOLLOWING PROGRESSION ON FIRST LINE CDK 4/6 INHIBITORAND AROMATASE INHIBITOR (FINER)

CCTG Protocol Number: MA.40

Prepared by:

Protocol Statistician: Bingshu Chen

Senior Investigator: Wendy Parulekar

Study Coordinator: Lisa Gallinaro

Study Chair: Stephan Chia

Date: February 15, 2025

 Doc. No.:
 MA.40

 Version:
 V001

 Date:
 2025-02-15

| Table of Con | | 2 |
|---|---|---|
| | n: | |
| • | ectives | |
| | ple Size Determination | |
| | ing of the Analyses | |
| | a Collection | |
| | nd Analyses | |
| | lyses Samples | |
| | ventions for Calculating Key Data | |
| | lysis Conventions | |
| | domization and Pre-treatment Characteristics | |
| 2.4.1 D | efinitions and Variables | |
| 2.4.1.1 | Accrual | |
| 2.4.1.2 | Randomization/Stratification | 5 |
| 2.4.1.3 | Ineligibility and Major Protocol Violations | 5 |
| 2.4.1.4 | Summary of Follow-up | 5 |
| 2.4.1.5 | Patient Characteristics | 6 |
| 2.4.1.6 | Baseline Cancer Treatment | 6 |
| 2.4.1.7 | Baseline Hematology/Biochemistry | 6 |
| 2.4.1.8 | Baseline Non-Hematologic Adverse Events | 7 |
| 2.4.2 Aı | nalysis of pre-treatment characteristics | 7 |
| 2.5 Effic | cacy | 7 |
| 2.5.1 D | efinitions and Variables | 7 |
| 2.5.1.1 | Progression-free Survival (PSF) | 7 |
| 2.5.1.2 | Overall Survival (OS) | 8 |
| 2.5.1.3 | Response rate | 8 |
| 2.5.1.4 | Duration of the response | 8 |
| 2.5.1.5 | Clinical benefit rate | 8 |
| 2.5.1.6 | Time to commencement of subsequent line of systemic therapy or death (TSST) | 8 |
| 2.5.2 Aı | nalysis of Key Parameters | 8 |
| 2.5.2.1 | Progression-free Survival | 9 |
| 2.5.2.2 | Overall Survival, TSST | 9 |
| 2.5.2.3 | Response rate and clinical benefit rate | 9 |
| 2.6 Dru | g Exposure | 9 |
| | -<br>rty | |
| 2.7.1 D | efinitions and Variables | 10 |
| 2.7.1.1 | Non-hematologic adverse events | 10 |
| 2.7.1.2 | Hematology/Biochemistry | |
| 2.7.1.3 | Serious adverse event | |
| 2.8 Off- | study and death | |
| | lity of Life | |
| | efinitions and Variables | |
| | EORTC QLQ-C30 | |
| | nalysis | |
| | Determination of Assessment Times | |
| | Calculation of Compliance Rates | |

# Statistical Analysis Plan (SAP)

 Doc. No.:
 MA.40

 Version:
 V001

 Date:
 2025-02-15

| | 2.9.2.3 Cross-sectional analysis | 13 |
|---|---|---|
| | 2.9.2.4 QOL response analysis | 13 |
| | 2.9.2.5 QOL subscale trend analysis | 13 |
| 3 Tal | bles | |
| | Table 1 Accrual by centre | 15 |
| | Table 2: Accrual by Stratification Factors at Randomization | 15 |
| | Table 3: Treatment received | 16 |
| | Table 4: Stratification factor at randomization vs. at baseline | 17 |
| | Table 5: Eligibility status | 18 |
| | Table 6: Summary of Follow-up | 18 |
| | Table 7: Patient characteristics | 19 |
| | Table 8. Baseline Hematology / Biochemistry | 20 |
| | Table 9. Baseline Non-Hematologic Adverse Event | 20 |
| | Table 10. Log Rank and Cox Regression Model for PFS Survival | 21 |
| | Table 11: PFS by Subsets | 22 |
| | Table 12: PFS Event Summary | 23 |
| | Table 13. Log Rank and Cox Regression Model for Overall Survival | 24 |
| | Table 14: OS by Subsets | 25 |
| | Table 15: Death Summary | 26 |
| | Table 16. Best response | 27 |
| | Table 16a. Response duration | 27 |
| | Table 17. Drug exposure | 27 |
| | Table 18. Non-Hematology adverse events | 28 |
| | Table 19. Hematology / Biochemistry (Follow-up) | 28 |
| | Table 20. Serious Adverse Events | 28 |
| | Table 21. Off protocol treatment | 28 |
| | Table 22. Death on Trial within 30 days of last treatment | 29 |
| | Table 23. Dates used to derive the Last know alive date (LKAD) | 30 |
| | Figure 1. KM plot for PFS | 31 |
| | Figure 2. KM plot for OS | 31 |
| | Figure 3. KM plot for Duration of response | 31 |
| | Figure 4. KM plot for TSST | 31 |

Doc. No.: MA.40 Version: V001

Date: 2025-02-15

#### 1 Introduction:

MA.40 is an international multi-centre, double-blind, randomized phase III trial comparing ipatasertib and fulvestrant with placebo and fulvestrant in patients with advanced (metastatic or loco-regionally recurrent not amenable to curative therapy) estrogen receptor positive (ER+) and human epidermal growth factor receptor 2 (HER-2) negative breast cancer after progression on first-line CDK 4/6 inhibitor and aromatase inhibitor (AI). This document describes the statistical analysis plan for the final analysis of MA.40.

#### 1.1 Objectives

The Primary Objective of the trial is to compare investigator-assessed progression-free survival (PFS) using RECIST 1.1 in patients with ER+/HER2- advanced (metastatic or loco-regionally recurrent not amenable to curative therapy) breast cancer treated with ipatasertib and fulvestrant versus placebo and fulvestrant after progression on first-line CDK 4/6 inhibitor plus AI treatment. The key Secondary Objective is to compare PFS by RECIST 1.1 in the PIK3CA/AKT1/PTEN altered cohort. Other secondary objectives include comparing the following endpoints: PFS by RECIST 1.1 in the PIK3CA/AKT1/PTEN altered cohort, PFS by central radiology review, Response Rate by RECIST 1.1, Duration of response, Clinical benefit rate, Overall Survival (OS), Time to commencement of subsequent line of systemic therapy or death (TSST), adverse events, health-related quality of life and health economic.

### 1.2 Sample Size Determination

The statistical assumptions for the control arm are based on the median PFS of 4.8 months in the control arm of FAKTION (though no prior CDK 4/6 inhibitor exposure in this trial) and the median PFS of 5.6 months in the control arm of SOLAR-1 (6% prior CDK 4/6 inhibitor exposure). Thus we assume an H0 median PFS of 4.5 months for the placebo + fulvestrant arm. Assuming a projected hazard ratio (HR) of 0.60 of benefit and thus a projected median PFS of 7.5 months in the ipatasertib and fulvestrant arm (H1 median PFS of 7.5 months) with an  $\alpha$  = 0.05 (2-sided) and 92% power, a total of 250 randomized patients (ITT population) will be required. The enrollment duration will be 24 months with 30 additional months for follow-up for the secondary and overall survival endpoints. 175 events will be required to trigger the final analysis for PFS. If PFS is significant for the ITT population at 0.05 level, then the pre-specified secondary analysis for the altered subgroup will be conducted. Assuming that the incidence rate of mutations is 45% and two-sided alpha = 0.05, the power to detect a hazard ratio of 0.50 (median PFS 3.5 months versus 7.0 months) will be 87% with a total of 79 PFS events.

For the secondary endpoint of OS, it is estimated that 76 deaths will have occurred at the time of the final PFS analysis. This will provide 34% power to establish an OS benefit with an HR of 0.70 for the OS endpoint. This projection is based on an estimated median OS in the control arm of 30 months and a projected median OS of 42.86 months in the ipatasertib + fulvestrant arm.

An additional OS analysis is planned when 155 deaths are observed. This will provide 60% power to establish an OS benefit with an assumed HR of 0.70 for OS (duration of follow-up of 30 months). These projections are based on an estimated median OS in the control arm of 30 months and a projected median OS of 42.86 months in the ipatasertib + fulvestrant arm.

### 1.3 Timing of the Analyses

The clinical cut-off date for this final analysis was June 4th, 2024. The database will be locked for on xxxx xxth, 2025 for the analysis.

#### 1.4 Data Collection

Data are collected, entered and managed by CCTG, Kingston, Ontario, according to the group standard data management procedure.

## 2 Methods and Analyses

### 2.1 Analyses Samples

The study populations for this analysis will include both the intention to treat (ITT) and as treated populations with data included as specified by the data cutoff date.

Analysis of pretreatment characteristics and all efficacy outcomes such as PFS and OS, will be based on the ITT population. A sensitivity analysis for efficacy outcomes will be conducted for the treated population. Those who received at least one dose of protocol therapy (i.e. the as-treated population) will form the basis of the safety analyses. The efficacy data set consists of all patients regardless of actual treatment.

### 2.2 Conventions for Calculating Key Data

In general, baseline evaluations are those collected closest, but before or on the day of randomization. If the pre-randomization assessment was not done, a pre-treatment assessment will be used as baseline assessment.

When either the day or month of a date is missing, the missing day or month will be imputed by the midpoints within the smallest known interval. For example, if the day of the month is missing for any date used in a calculation, the 15th of the month will be used to replace the missing day. If the month and day of the year are missing for any date used in a calculation, the first of July of the year will be used to replace the missing data. The partial date imputation will be applied to adverse event (AE) start date and concomitant medication (CM) start date only.

### 2.3 Analysis Conventions

When converting a number of days to other units, the following conversion factors will be used:

1 year = 365.25 days

1 month = 30.4375 days

All comparisons between treatment arms will be carried out using a two-sided test at an alpha level of 5% unless otherwise specified. No formal adjustments will be made for the multiplicity of inferences for the other clinical endpoints.

Date. 2020-02-10

The following baseline stratification factors that will be used to adjust the analyses where appropriate are listed below:

- PIK3CA/PTEN/AKT1 alteration status: altered versus wildtype/unknown
- Prior duration of treatment with CDK 4/6 inhibitor: < 6 months versus ≥ 6 months</li>

## 2.4 Randomization and Pre-treatment Characteristics

## 2.4.1 Definitions and Variables

## 2.4.1.1 Accrual

• Number (%) of randomized patients per study center and country (table 1). This table is for CCTG internal use only.

## 2.4.1.2 Randomization/Stratification

- PIK3CA/PTEN/AKT1 alteration status: altered versus wildtype/unknown
- Prior duration of treatment with CDK 4/6 inhibitor: < 6 months versus ≥ 6 months</li>
- Centre: was used as a stratification factor in the randomization but will not be used in the stratified analysis

A minimization procedure for treatment assignment was used in this study. Stratification factors at randomization will be summarized by the treatment arm (table 2).

The number and percentage of actual treatment received will be summarized by arm (table 3).

Treatment at randomization will be compared with the actual treatment received to identify any discrepancies (table 4).

## 2.4.1.3 Ineligibility and Major Protocol Violations

The number and percentage of ineligible patients will be presented by the treatment arm.

Reasons for ineligibility: The percentage for each reason and combination of reasons of ineligibility will be presented by the treatment arm.

The number and percentage of major protocol violations will be presented by the treatment arm (table 5).

### 2.4.1.4 Summary of Follow-up

<sup>\*</sup>Add missing/unknown category whenever appropriate.

## Statistical Analysis Plan (SAP)

Doc. No.: MA.40 Version: V001 Date: 2025-02-15

A table showing the median, min and max follow-up (defined as reverse censoring on overall survival) will be presented by treatment group and for all patients included in the analysis (table 6).

#### 2.4.1.5 Patient Characteristics

Patient characteristics at baseline are summarized in table 7.

- Age
- Sex
- BMI
- Race
- ECOG PS
- ER status: Positive VS Negative (all patients shall be ER positive)
- PR status: Positive VS Negative
- HER2 status: 0, 1,2, 3 (all patients shall be HER 2 negative)
- Stage IV at diagnosis (Yes vs No)
- Site of disease
  - Sites of disease < 3 versus > or = 3
  - o Bone only
  - Liver involvement
  - Lung involvement
  - Lung or liver involvement

### 2.4.1.6 Baseline Cancer Treatment

The number and percent of patients who received cancer treatment (Chemotherapy, Hormone Therapy (Neoadj vs post op), Immunotherapy, Adjuvant therapy, Neo-adjuvant therapy, Radiotherapy, Other therapy) will be summarized by treatment arm (table 7).

## 2.4.1.7 Baseline Hematology/Biochemistry

CTC 4.0 grades will be used to summarize the baseline hematology/biochemistry data (% with each CTC grade) for the following assessments (table 8):

- WBC,
- Granulocytes,
- Platelets,
- Hemoglobin
- Bili
- AST, ALT,
- Alk phosph
- Glucose

- HgAlc
- Albumin
- Creatinine

#### 2.4.1.8 Baseline Non-Hematologic Adverse Events

CTC V 5.0 grades will be used to summarize the baseline non-hematologic (number for each CTC grade, total number and %) (table 9).

#### 2.4.2 Analysis of pre-treatment characteristics

No formal statistical tests will be performed to assess the homogeneity of baseline characteristics between the arms. Categorical variables will be tabulated by the treatment arm and for all patients. Continuous variables (e.g., age) or transformed continuous variables will be presented using summary statistics (n, mean, standard deviation (SD), median, min and max) or specified cutoff categories by treatment arm and for all patients. Analyses will be based on all randomized patients by arm based on the ITT population.

#### 2.5 Efficacy

## 2.5.1 Definitions and Variables

#### 2.5.1.1 Progression-free Survival (PFS)

The primary endpoint is progression-free survival (PFS) defined as time from randomization to disease progression or death from any cause, whichever occurs first. Disease progression will be investigator-assessed using the RECIST 1.1 criteria. CCTG or its designee will collect and store all tumour measurement images on all enrolled patients throughout the study to enable an independent review of imaging scans and an assessment of disease progression. If a patient has not progressed or died at the time of final analysis, PFS will be censored on the date of the last visit with adequate disease assessment. Lack of tumour assessments post-randomization or leak of baseline assessment will lead to censoring on day one after randomization. Progression documented between scheduled visits will be assigned to the date of the clinical lesion evaluation indicating progression. Death before the first PD assessment, including death between adequate assessment visits, will lead to the assignment of progression to the date of death. Death or progression after more than one missed visit will lead to the censoring of data at the date of the last visit with adequate assessment. Patients who received non-protocol anti-cancer treatment prior to a PFS event will be censored at the date of commencement of the non-protocol anti-cancer treatment.

## PFS Time (months) =

((date of PFS event or last disease assessment date - date of randomization) + 1) / 30.4375

### 2.5.1.2 Overall Survival (OS)

For patients who have died, overall survival is calculated in months from the day of randomization to the date of death. Otherwise, survival is censored on the last day the patient is known alive date (LKAD).

OS Time (months) = ((date of death or LKAD - date of randomization) + 1) / 30.4375

Where the LKAD is defined in Table 23.

#### 2.5.1.3 Response rate

Response rate (RR) per RECIST 1.1 is defined as the number of responders (complete response and partial response, non-CR/PR for patients without measurable disease)) as a percentage of all the randomized patients.

## 2.5.1.4 Duration of the response

Duration of Response (DoR) will be calculated for patients with an overall best response of CR or PR as per RECIST 1.1 criteria. DoR is measured from the date of first evidence of CR or PR to the date of objective progression or the date of death due to any cause, whichever is earlier. If a patient has not progressed or died at the time of the final analysis, the duration of response will be censored on the date of the last disease assessment.

### 2.5.1.5 Clinical Benefit Rate

Clinical Benefit Rate (CBR) will be calculated for the number of patients with an overall best response of CR, PR or SD ( $\geq$  6 months) as per RECIST 1.1 criteria as a percentage of all randomized patients. SD duration greater or equal to 6 months is defined as the date of randomization to the earliest of the date of objective progression, the date of death due to any cause, or the date of last disease assessment is greater or equal to 6 months.

## 2.5.1.6 Time to Commencement of Subsequent Line of Systemic Therapy or Death (TSST)

Time to commencement of subsequent line of systemic therapy or death (TSST) is defined as the time from randomization to the time of subsequent treatment commencement or death, whichever comes first. TSST will be censored at the date of last known alive without commencement of subsequent line of systemic therapy.

## 2.5.2 Analysis of Key Parameters

The comparison between treatment arms will be carried out using a two-sided test at an alpha level of 5% unless otherwise specified. All efficacy analyses will be presented by the treatment arm. The CONSORT diagram will be included.

## 2.5.2.1 Progression-free Survival

The primary PFS comparison between treatment arms will be performed on data derived from the ITT population. All patients will be included in the primary PFS efficacy analyses according to the arm of randomization, regardless of the actual treatment received. The PFS survival experiences of subjects in both treatment arms will be described by the Kaplan-Meier method. Stratified two-sided log-rank tests adjusting for stratification factors as defined in the protocol will be the primary method to compare PFS between the experimental and control arms. As an exploratory analysis, a Cox proportional hazards model will be used to identify and adjust for factors significantly related to progression-free survival.

A pre-specified secondary analysis for PFS in the PIK3CA/PTEN/AKT1 altered status subset will be tested using a hierarchical testing procedure [Hung, 2007]. If the result for PFS in the ITT patient population is significant at a 0.05 level, then PFS will be tested in the PIK3CA/PTEN/AKT1 altered status subset under the same 0.05 significance level. If this criterion for the PFS comparison is not met in the ITT population, no further testing for the PFS comparison will be performed in the PIK3CA/PTEN/AKT1 altered status subgroup. (Table 10, 11, Figure 1).

For patients who developed PFS events, the type of progression events and summary of progression will be tabulated (Table 12).

As a pre-specified secondary analysis, PFS analysis will be repeated by PFS events based on central radiology review.

#### 2.5.2.2 Overall Survival, TSST

The analyses of OS and TSST will be similar to these of PFS (Table 13, 14, 15, Figure 2, 4).

## 2.5.2.3 Response Rate and Clinical Benefit Rate

The number and percentage of CR, PR, SD, and PD will be reported (Table 16).

The 95% confidence intervals for the response rate and clinical benefit rate will be calculated for each arm. The difference in response rate between the two arms and the corresponding 95% confidence interval will be obtained by the asymptotic normal approximation.

Median for the duration of the response will be calculated using the KM method for each arm (Table 16a).

#### 2.6 Drug Exposure

Duration of drug exposure (fulvestrant and ipatasertib / placebo) will be reported as time from the date of the first dose of protocol therapy to the time of the last drug dose before the clinical cut-off date. The date of randomization will be used if the first dose date is unknown. If the date of discontinuation is

## Statistical Analysis Plan (SAP)

Doc. No.: MA.40 Version: V001 Date: 2025-02-15

unknown, we use the drug injection date for fulvestrant and the drug start date + 21 days for ipatasertib / placebo.

The min, median, mean, standard deviation, and max duration of drug exposure will be reported by the treatment arm in Table 17.

#### 2.7 Safety

## 2.7.1 Definitions and Variables

All toxicity/side effects data collected post-randomization will be included in the analyses of toxicities.

#### 2.7.1.1 Non-hematologic Adverse Events

Non-hematologic adverse events will be summarized according to CTC AE 5.0 (Table 18).

## The number and percentage for Adverse Events of Special Interest (AESI) will be reported.

- Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's law.
- Grade ≥ 3 hepatotoxicity.
- Grade ≥ 3 ALT/AST elevations.
- Suspected transmission of an infectious agent by the study drug, defined as any organism, virus
  or infectious particle (e.g. prion protein transmitting/transmissible spongiform encephalopathy),
  pathogenic or non-pathogenic, is considered an infectious agent. A transmission of an infectious
  agent may be suspected from clinical symptoms or laboratory findings that indicate an infection
  in a patient exposed to a medicinal product. This term applies only when a contamination of the
  study drug is suspected.
- Grade ≥ 3 diarrhea.
- Grade ≥ 3 fasting hyperglycemia.
- Grade ≥ 2 pneumonitis.
- Grade ≥ 2 colitis/enterocolitis.
- Grade ≥ 3 rash.
- Erythema multiforme

## 2.7.1.2 Hematology/Biochemistry

Hematology/Biochemistry experience will be reported according to CTC AE 5.0 (Table 19).

## 2.7.1.3 Serious Adverse Event

SAE will be listed by treatment arm (Table 20).

#### 2.8 Off-study and Death

Patients off-study (off protocol treatment): Number and % of all treated patients. Reason for going off-study (e.g. adverse event, death, progression, etc.): The number and % of all treated patients will be presented (table 21).

Deaths within 30 days from the last treatment administration. Cause of death within 30 days from the last treatment administration: The number and % of all treated patients will be presented (table 22).

## 2.9 Quality of Life

The EORTC QLQ-C 30 Global Score will be used for our primary assessment of quality of life.

#### 2.9.1 Definitions and Variables

#### 2.9.1.1. EORTC QLQ-C30

There are five functional domains and three symptom domains that can be derived from EORTC QLQ-C30 (see below for definitions). If the number of unanswered questions in each domain is within a limit specified with the definition for each domain, the score is calculated as below:

#### For function domains of Physical, Emotional, Cognitive and Social:

Score = 100-(((Total score for the answered questions / (Total questions answered))-1)\*100/3).

#### For symptom domains:

Score = (((Total for the answered questions / (Total questions answered))-1)\*100/3)

Otherwise, the score will be recorded as "missing". For each single item, the score will be recorded as "missing" if the answer to this item is missing.

### **Functional Domains:**

Physical: Questions: 1, 2, 3, 4, 5

Score=missing if the number of above questions not answered is greater than 2;

Role: Questions: 6, 7

Score=missing if the number of above questions not answered is greater than 1;

Emotional: Questions: 21, 22, 23, 24

Score=missing if the number of above questions not answered is greater than 2;

Cognitive: Questions: 20, 25

Score=missing if the number of above questions not answered is greater than 1;

Social: Questions: 26, 27

Score=missing if the number of above questions not answered is greater than 1;

## **Symptom Domains:**

Fatigue: Questions: 10, 12, 18

Score=missing if the number of above questions not answered is greater than 1;

Nausea and vomiting: Questions: 14, 15

Score=missing if the number of above questions not answered is greater than 1;

Pain: Questions: 9, 19

Score=missing if the number of above questions not answered is greater than 1.

There are also six single items in EORTC QLQ-C30 about common symptoms and one global assessment that can be derived from EORTC QLQ-C30. The single items are:

## Single Items:

Dyspnea: Question 8;
Sleep/Insomnia: Question 11;
Appetite: Question 13;
Constipation: Question 16;
Diarrhea: Question 17;
Financial: Question 28.

They are all scored using the following formula:

Score= (Answer to the question-1)\*100/3.

The Global Assessment includes Questions 29 and 30. If number of the questions not answered is greater than 0, its score will be "missing"; Otherwise,

Score= ((Total for the answered questions / (Total questions answered))-1)\*100/6.

For functional domains, a higher score indicates better functioning but for symptom domains, a higher score indicates higher (worse) symptoms.

#### 2.9.2 Analysis

All analyses on quality of life scores will be exploratory and will **include all randomized patients with QOL data**.

#### 2.9.2.1 Determination of Assessment Times

The following will be the scheme to determining the time frame of a QOL assessment:

- 1) Baseline: Baseline evaluation is the QOL questionnaire collected closest, but prior to, the first day of starting study treatment/randomization;
- 2) Day 1 of cycle 2: If the QOL is assessed between days -2 to 27 of cycle 2
- 3) Day 1 of cycle 3: If the QOL is assessed between days -2 to 27 of cycle 3
- 4) Day 1 of cycle 4: If the QOL is assessed between days -2 to 27 of cycle 4
- 5) Cycle 5, 7, 9, 11: If the QoL is assessed between days 2 to 27 of cycle 5, 7, 9, 11.
- 6) 4 weeks after complete of protocol treatment: If the QOL is assessed between weeks 2 and 8 after the protocol treatment

Doc. No.: MA.40 Version: V001

Date: 2025-02-15

### 2.9.2.2 Calculation of Compliance Rates

The following method will be used to calculate the compliance rates of QOL assessment. The compliance rate is calculated as the number of forms received out of the number of forms expected at each assessment point defined based on the following principles:

- 1) At baseline: the number of forms expected is the total number of patients who are required to fill out QOL questionnaires.
- 2) FU period: the number expected at each assessment is the number of patients with baseline data minus the number of patients who have died or progressed during that and previous follow-up period (with assessment window defined by 2.9.2.1).

#### 2.9.2.3 Cross-sectional Analysis

The mean and standard deviation of QOL scores at baseline and the mean and standard deviation of QOL change scores from baseline at each assessment time will be calculated. Then Wilcoxon Rank-Sum test is used to compare two treatment arms in terms of change in QOL score at each assessment time from baseline.

Mean change in scores over time will be analyzed using a generalized linear mixed model. The treatment arms and QOL assessment time points will be used as covariates in this analysis. The interactions between treatment arms and QOL assessment time (baseline to week 4 after treatment) will be tested using a likelihood ratio method.

#### 2.9.2.4 QOL Response Analysis

QOL response is calculated as follows for a functional domain: A change score of 10 points from baseline was defined as clinically relevant. Patients will be assessed as improved if they have reported a score of 10 points or better than baseline at any time of the QOL assessment. Conversely, patients will be assessed as worsened if there is a reported score that is at least 10 points worse than baseline at any time of the QOL assessments without meeting the criteria for improvement. Patients whose scores are intermediate between these values at every QOL assessment will be considered as stable. In contrast to functional domains, for the determination of a patient's QOL response, the classification of patients into improved and worsened categories is reversed for symptom domains and single items. A Chi-square test will be performed to compare the distributions of these three categories between two arms (improved, stable or worse).

#### 2.9.2.5 QOL Subscale Trend Analysis

Plots of QoL scores over time by treatment arms over time (From baseline to week 4 after treatment) will be reported for global QOL, each subscale and symptom item.

Note: Patient-reported outcomes version of the adverse events (PRO-CTCAE), health economic and correlative sciences will be analyzed separately.

## 3 Tables

## Table 1 Accrual by Centre

| Centre | 1 | Number of accrual (%) | |
|--------|------------------------|-----------------------|------------------|
| | Ipatasertib<br>N = *** | Placebo<br>N = *** | Total<br>N = *** |
| Xxxx | XX (XX) | XX (XX) | XX (XX) |

Table 2: Accrual by Stratification Factors at Randomization

| | Data set: All Rando | omized Patients | |
|---|---|---|---|
| | Number of patients (%) | | |
| | Ipatasertib<br>N = *** | Placebo<br>N = *** | Total<br>N = *** |
| PIK3CA/PTEN/AKT1 | | | |
| Altered | ** (**) | ** (**) | ** (**) |
| Wildtype/Unknown | ** (**) | ** (**) | ** (**) |
| Prior duration of treatment with CDK 4/6 inhibitor | | | |
| <6months | | | |
| >/=6months | ** (**) | ** (**) | ** (**) |
| | ** (**) | ** (**) | ** (**) |
| Source: Centralized Rand | omization File | | |

Doc. No.: MA.40 V001 2025-02-15 Version:

Date:

## **Table 3: Treatment Received**

| Number of accrual (%) | | |
|---|---|---|
| Ipatasertib<br>N = *** | Placebo<br>N = *** | Total<br>N = *** |
| XX (XX) | XX (XX) | XX (XX) |
| | Ipatasertib<br>N = *** | Ipatasertib Placebo N = *** N = *** |

<u>Table 4: Stratification Factor at Randomization vs. at Baseline</u>

| | Data set: All Rando | mized Patients | |
|---|---|---|---|
| | Number of patients (%) | | |
| At randomization | At baseline | Ipatasertib<br>N = *** | Placebo<br>N = *** |
| PIK3CA/PTEN/AKT1 | | | |
| Altered | Altered | ** (**) | ** (**) |
| Wildtype/Unknown | Altered | ** (**) | ** (**) |
| Altered | Wildtype/Unknown | | |
| Wildtype/Unknown | Wildtype/Unknown | | |
| Prior duration of treatment with CDK 4/6 inhibitor | | ** (**) | ** (**) |
| <6months | <6months | ** (**) | ** (**) |
| >/=6months | <6months | | |
| <6months | >/=6months | | |
| >/=6months | >/=6months | | |

**Table 5: Eligibility Status** 

| Total patients allocated | Ipatasertib | Placebo | Total |
|---------------------------|-------------|---------|---------|
| | N = *** | N = *** | N = *** |
| Ineligible | XX (XX) | | |
| Total eligible patients | XX (XX) | | |
| REASONS FOR INELIGIBILITY | | | |
| Reason 1 | XX (XX) | | |
| Reason 2 | XX (XX) | | |
| Major Protocol Violations | | | |
| XXX | | | |
| XXX | | | |

Table 6: Summary of Follow-up

| Data set: All Randomized Patients | | | |
|---|---|---|---|
| | | Number of patients | |
| | Placebo<br>N = *** | · | |
| Median* | *** | *** | *** |
| Min | ** | ** | ** |
| Max | ** | ** | ** |

Median Follow-up based on inverse OS

## <u>Table 7: Patient Characteristics</u>

| All randomized patients | Ipatasertib<br>N = *** | Placebo<br>N = *** | Total<br>N = *** |
|---|---|---|---|
| AGE | | | |
| <=39 | XX (XX) | | |
| 40-49 | XX (XX) | | |
| 50-59 | , | | |
| 60-69 | | | |
| >=70 | XX (XX) | | |
| Median (Range) | XX (XX) | | |
| Sex | | | |
| M | | | |
| F | | | |
| Race | | | |
| Ethnicity | | | |
| ECOG PS | | | |
| 0 | | | |
| 1 | | | |
| 2 | | | |
| Prior Chemotherapy in advanced disease setting (Y versus N) | | | |
| Sites of metastases <3 Or =3 | | | |
| Bone only | | | |
| Lung involvement | | | |
| Liver involvement | | | |
| Lung or Liver involvement | | | |
| Tang or Liver involvement | | | |
| ER status | | | |
| Positive | | | |
| Negative | | | |
| PR status | | | |
| Positive | | | |
| Negative | | | |
| HER2 status | | | |
| 11ENZ Status | | | |

# Statistical Analysis Plan (SAP)

Doc. No.: MA.40 Version: V001 Date: 2025-02-15

| 1 |
|---|
| 2 |
| 3 |

Table 8. Baseline Hematology / Biochemistry

CTC AE 5.0 Hematology / Biochemistry table

<u>Table 9. Baseline Non-Hematologic Adverse Events</u>

CTC AE 5.0 Non-Hematologic Adverse Event table

Table 10. Log Rank and Cox Regression Model for PFS Survival

| Data set: | All Randomized | d Patients | | |
|---|---|---|---|---|
| | Univariate | Log-rank | Multivariate | Multivariate |
| | HR (95% CI) | p-value | HR(95% CI) (1) | p-value |
| Treatment (Ipatasertib vs. Placebo) (stratified at randomiation) | *** | *** | | |
| Treatment (Ipatasertib vs. Placebo) (un-stratified) | | | | |

<sup>(1)</sup> Based on the Cox Model with all factors included.

 Doc. No.:
 MA.40

 Version:
 V001

 Date:
 2025-02-15

## Table 11: PFS by Subsets

| | Data set: All Rand | | |
|---|---|---|---|
| | | Number of patients (%) | |
| | Ipatasertib | Placebo | HR |
| | N (# of event) | N (# of event) | (95% C.I) |
| PIK3CA/PTEN/AKT1 | | | |
| Altered | ** (**) | ** (**) | (**, **) |
| Wildtype/Unknown | ** (**) | ** (**) | (**,**) |
| Prior duration of treatment with CDK | | | |
| 4/6 inhibitor<br><6months | ** (**) | ** (**) | (**,**) |
| >/=6months | ** (**) | ** (**) | (**,**) |

## **Table 12: PFS Event Summary**

| | domized Patients Number of Patients (%) | |
|---|---|---|
| | Ipatasertib | Placebo |
| | N = *** | N = *** |
| Patients with PFS event | *** (**) | *** (**) |
| Progression | ** | ** |
| <u> </u> | ** | ** |
| | ** | ** |
| | ** | ** |
| | ** | ** |
| | ** | ** |
| | ** | ** |
| Death | ** | ** |
| Patients who were censored | *** (**) | *** (**) |
| Reason Censored | . , | |
| No PFS event | ** | ** |
| Withdrawal of Consent | ** | ** |

Table 13. Log Rank and Cox Regression Model for Overall Survival

| Data set: All Randomized Patients | | | | |
|---|---|---|---|---|
| | Univariate<br>HR (95% CI) | Log-rank<br>p-value | Multivariate<br>HR(95% CI) <sup>(1)</sup> | Multivariate<br>p-value |
| Treatment (Ipatasertib vs. Placebo) (stratified) | *** (*, *) | *** | *** (*, *) | *** |
| Treatment (Ipatasertib vs. Placebo) (un-stratified) | *** (*, *) | *** | *** (*, *) | *** |
| | *** (*, *) | *** | *** (*, *) | *** |
| | *** (*, *) | *** | *** (*, *) | *** |
| | *** (*, *) | *** | *** (*, *) | *** |
| Other factors | | | | |

(1) Based on the Cox Model with all factors included.

.

 Doc. No.:
 MA.40

 Version:
 V001

 Date:
 2025-02-15

## Table 14: OS by Subsets

| | Data set: All Rand | omized Patients | |
|---|---|---|---|
| | | Number of patients (%) | |
| | Ipatasertib | Placebo | HR |
| | N (# of event) | N (# of event) | (95% C.I) |
| PIK3CA/PTEN/AKT1 | | | |
| Altered | ** (**) | ** (**) | (** , **) |
| Wildtype/Unknown | ** (**) | ** (**) | (** , **) |
| Prior duration of | | | |
| treatment with CDK 4/6 inhibitor | | | |
| <6months | ** (**) | ** (**) | (**, **) |
| >/=6months | ** (**) | ** (**) | (**,**) |

 Doc. No.:
 MA.40

 Version:
 V001

 Date:
 2025-02-15

Table 15: Death Summary

| | Number of Patients (%) | | |
|---|---|---|---|
| | Data set: All randomized Patients | | |
| | Ipatasertib | Placebo | Total |
| | N = | N = | N = |
| Patients who died | | | |
| Cause of Death | | | |
| Breast Cancer only | | | |
| Other primary malignancy | | | |
| Other conditions or | | | |
| circumstances | | | |
| Patients who were censored | | | |
| Reason Censored | | | |
| Still Alive | | | |
| Withdrawal of Consent | | | |

## Table 16. Best Response

| | Data set: All Rand | domized Patients | |
|---|---|---|---|
| | Number of patients | | |
| | Placebo Ipatasertib Total N = *** N = *** N = *** | | |
| CR | XX (%) | XX (%) | XX (%) |
| PR | ** | ** | ** |
| SD | ** | ** | ** |
| PD | | | |
| In-evaluable | | | |

## Table 16a. Response Duration

| | Data set: All Rand | omized Patients | |
|---|---|---|---|
| | Number of patients | | |
| | Placebo Ipatasertib Total N = *** N = *** N = *** | | |
| Median* | *** | *** | *** |
| Min | ** | ** | ** |
| Max | ** | ** | ** |

<sup>\*</sup> Based on the KM method

Table 17. Drug Exposure

| Data set: All treated Patients | | | |
|---|---|---|---|
| | Number of patients | | |
| | Placebo | Placebo Ipatasertib Total N = *** N = *** N = *** | |
| | N = *** | N = *** | N = *** |
| Median* | *** | *** | *** |
| Min | ** | ** | ** |
| Max | ** | ** | ** |

## <u>Table 18. Non-Hematologic Adverse Events</u>

CTC AE 5.0 non-hematology adverse events table

## Table 19. Hematology / Biochemistry (Follow-up)

CTC AE 5.0 Hematology / Biochemistry table

## Table 20. Serious Adverse Events

As in the meeting book table.

Table 21. Off Protocol Treatment

| | Data set: All tr | eated Patients | |
|---|---|---|---|
| | Number of patients | | |
| Off treatment | Ipatasertib<br>N = *** | Placebo<br>N = *** | Total<br>N = *** |
| Cause1 | *** | *** | *** |
| 2 | ** | ** | ** |
| 3 | | | |
| 4 | | | |

Note: One table for each type of treatment (oral and iv)

<u>Table 22. Death on Trial within 30 days of last Treatment</u>

| | Data set: All tre | eated Patients | |
|---|---|---|---|
| | Number of patients | | |
| Cause of Death | Ipatasertib<br>N = *** | Placebo<br>N = *** | Total<br>N = *** |
| Cause1 | *** | *** | *** |
| 2 | ** | ** | ** |
| 3 | | | |
| 4 | | | |

Table 23. Dates Used to Derive the Last Known Alive date (LKAD)

| CDASH data | CRF Section | Date Variable as the source of | Description | Note |
|---|---|---|---|---|
| | Name | LKAD | | |
| MA40_WC | Withdraw of | DS_DSSTDAT_ | Date of consent withdrawal | |
| | consent | WITHDRAWAL | | |
| MA40_LTFU | Lost to follow-up | DS_DSSTDAT_LOST | Date of lost to follow-up | |
| MA40_F5 MA40_F5P | Form 5/ Form 5s/ | VISDAT | End date of visit | |
| MA40_F5S | Form 5p | | | |
| MA40_F9 | F9 | RS_RSDAT | Date of Relapse / Progression | |
| MA40_PE | Physical Exam | VISDAT | Date of Exam | Post<br>baseline |
| MA40_TRT_IV | Drug<br>Administration | EC_ECSTDAT | Dose administrate date where the EC_ECDSTXT_PERFORMED (actual dose given) not equal to 0. | IM<br>protocol<br>therapy |
| MA40_LES_TAR | Lesion | TU_TUDAT | Date of Test for Target, non-target | Post |
| MA40_LES_NTAR | evaluation | | and new lesion | baseline |
| MA40_LES_NEW | | | | |
| MA40_RADIO | Other | TU_TUDAT_OTHERRAD | Assessment Date | Post |
| | Radiology<br>Investigations | | | baseline |
| MA40_LAB | Hematology and<br>Biochemistry | TEST_DT | Date of blood collection | Test<br>done |
| MA40_ECG | Cardiac<br>Function<br>( ECG) | EG_EGDAT | Date of ECG | Post<br>baseline |
| MA40_HOSP | Hospitalization | HO_HOSTDAT, HO_HOENDAT | Admission Date and Discharge Date | |
| MA40_AE | Adverse Event | AE_AESTDAT_PA, | Date of onset and Date of | complet |
| _ | (Post baseline<br>SAE only) | AE_AEENDAT_PA | Resolution of SAE only | e dates |
| MA40_LAB | Tests (Numeric) | TEST_DT | CollectionDate of Worst Value, | Post |
| | (SAE) | | Collection Date of recovery | baseline |
| MA40_SAE_NONNUM | Tests<br>(Nonnumeric)<br>(SAE) | STDAT_TESTS_SAE | Date of Test | |
| MA40_CANCERTX_1 | Cancer Treatment | PR_PRSTDAT_NEWTX_PA | date of surgery | complet |
| Treatment Folders only | (Surgery) | | | e dates |
| MA40_CANCERTX_2 | Cancer | PR_PRSTDAT_NEWTX_PA | First Fraction Date, | complet |
| Treatment Folders only | Treatment (RT) | PR_PRENDAT_NEWTX_PA | Last Fraction Date | e dates |
| MA40_CANCERTX_3 | Cancer Treatment | CM_CMSTDAT_NEWTX_PA, | Start Date | complet |
| Treatment Folders only | Systemic Therapy | CM_CMENDAT_PA | End Date | e dates |
| MA40_PREG | Pregnancy Test | LB_LBDAT_PREG | Date of pregnancy test | |

Figure 1. KM plot for PFS

Figure 2. KM plot for OS

Figure 3. KM plot for Duration of Response

Figure 4. KM plot for TSST